CLINICAL TRIAL: NCT01105585
Title: A Comparative Pilot Study Of High-Order Aberrations With Aspheric Intraocular Lens (IOL) Models SN60WF And ZCB00
Brief Title: A Comparative Pilot Study Of High-Order Aberrations With Aspheric IOL Models SN60WF and ZCB00
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: M-09-003
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Cataracts
Keywords: Cataracts; aspheric; IOL; ocular aberrations
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZCB00 IOL (Experimental): Tecnis 1-piece Aspheric Acrylic (ZCB00) intraocular lens (IOL) randomly assigned to one eye, with AcrySof Natural IQ (SN60WF) IOL in the fellow eye for contralateral implantation
  Interventions: Device: Tecnis 1-piece Aspheric Acrylic (ZCB00) IOL
- SN60WF IOL (Active Comparator): AcrySof Natural IQ (SN60WF) intraocular lens (IOL) randomly assigned to one eye, with Tecnis 1-piece Aspheric Acrylic (ZCB00) intraocular lens in the fellow eye for contralateral implantation
  Interventions: Device: AcrySof Natural IQ (SN60WF) IOL

INTERVENTIONS:
Device: Tecnis 1-piece Aspheric Acrylic (ZCB00) IOL — Tecnis 1-piece Aspheric Acrylic (ZCB00) intraocular lens implanted in the capsular bag during cataract surgery. The IOL is intended for the lifetime of the patient.
  Arms: ZCB00 IOL
Device: AcrySof Natural IQ (SN60WF) IOL — AcrySof Natural IQ (SN60WF) intraocular lens implanted in the capsular bag during cataract surgery. The IOL is intended for the lifetime of the patient.
  Arms: SN60WF IOL

SUMMARY:
The purpose of this study was to prospectively compare high-order aberrations between eyes implanted with the AcrySof® Natural IQ (SN60WF) intraocular lens (IOL) versus those implanted with the Tecnis ZCB00 IOL.

ELIGIBILITY:
Inclusion Criteria:

* Requires bilateral extraction of cataracts by phacoemulsification followed by implantation of a posterior chamber intraocular lens;
* Confirmed absence of pre-existing conditions that could skew the results or present contraindications for the IQ intraocular lens (IOL) or the Tecnis ZCB00 IOL;
* <1 diopter corneal astigmatism preoperatively;
* Able to achieve 6.5 mm dilated pupil;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Chronic disease or illness;
* Irregular optical aberration;
* Amblyopia;
* History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.);
* Diabetic retinopathy;
* Macular degeneration;
* History of retinal detachment;
* Other surgeries planned at time of cataract removal;
* Severe dry eye;
* Other protocol-defined exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Total ocular high-order aberrations | Month 1 postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States